CLINICAL TRIAL: NCT03784027
Title: Open-label, Multi-centre, Multi-national, Randomized 2-period Crossover Study Comparing Closed-loop Insulin Delivery With Sensor-augmented Pump Therapy Over 4 Months in Children 1-7 Years With Type 1 Diabetes at Home, With an Extension.
Brief Title: The Artificial Pancreas in Very Young Children With T1D
Acronym: KidsAP02
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: European Commission (Other); Cambridge University Hospitals NHS Foundation Trust (Other); The Leeds Teaching Hospitals NHS Trust (Other); University of Luxembourg (Other); University of Leipzig (Other); Medical University of Graz (Other); Medical University Innsbruck (Other); Medical University of Vienna (Other); Jaeb Center for Health Research (Other); University of Edinburgh (Other); Stanford University (Other); Glooko (Industry)
Responsible Party: Principal Investigator, Dr Roman Hovorka, Study Director, University of Cambridge
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KidsAP02
Record Dates: First submitted 2018-12-19; First posted 2018-12-21 (Actual); Results first posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Device: CamAPS FX
  The automated closed loop system (CamAPS FX) will consist of:
  * Dana RS insulin pump (Diabecare, Sooil, Seoul, South Korea)
  * Dexcom G6 real-time CGM sensor (Dexcom, Northridge, CA, USA)
  * An Android smartphone hosting CamAPS FX app with the Cambridge model predictive control algorithm and communicating wirelessly with the insulin pump and glucose sensor
  * Cloud upload system to monitor CGM/insulin data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Automated closed loop insulin delivery (intervention arm) (Experimental): Unsupervised home use of day and night automated hybrid closed loop insulin delivery system over 16 weeks.
  Intervention: Device: CamAPS FX
  Interventions: Device: CamAPS FX
- Sensor augmented pump therapy (control arm) (Active Comparator): Sensor augmented pump therapy over 16 weeks.
  Interventions: Other: Sensor augmented therapy

INTERVENTIONS:
Device: CamAPS FX — CamAPS FX closed loop system comprises:
  * Dana insulin pump (Diabecare, Sooil, Seoul, South Korea)
  * Dexcom G6 real-time CGM sensor (Dexcom, Northridge, CA, USA)
  * An Android smartphone hosting CamAPS FX app with the Cambridge model predictive control algorithm and communicating wirelessly with the insulin pump and glucose sensor
  * Cloud upload system to monitor CGM/insulin data
  Arms: Automated closed loop insulin delivery (intervention arm)
Other: Sensor augmented therapy — Study insulin pump and study CGM.
  Arms: Sensor augmented pump therapy (control arm)

SUMMARY:
The suggested clinical trial is part of the KidsAP project funded by the European Commission's Horizon 2020 Framework Programme and JDRF. It evaluates the use of the Artificial Pancreas (closed loop system) in very young children with type 1 diabetes (T1D) aged 1-7 years. This outcome study aims to determine whether 24/7 automated closed loop glucose control improves time in range compared to sensor augmented pump therapy. An extension phase will evaluate the effect of long-term home use of the 24/7 automated hybrid closed loop insulin delivery system on glucose control (UK sites only).

The study employs an open-label, multi-centre, multi-national, randomized, two-period, crossover design. Participants undergo a 2-4 week run-in period, followed by two 16-week treatment periods (one for each therapy) separated by a 1-4 week washout. The order of treatments is randomized. Up to 80 young children (with a target of 72 randomized subjects) on insulin pump therapy will be recruited from paediatric outpatient diabetes clinics.

Before using the study devices, participants and their parents/guardians receive training on the safe use of the study pump, continuous glucose monitoring (CGM) device, and hybrid closed loop system. Nursery or school carers may also be trained if needed. During the closed loop arm, subjects use the system for 16 weeks under free-living conditions at home and in nursery/school without remote monitoring. In the control arm, subjects use sensor augmented pump therapy for 16 weeks under similar conditions, with regular contact and 24/7 telephone support from the study team.

The primary endpoint is the time spent in the target glucose range (3.9-10.0 mmol/l) as recorded by CGM. Secondary outcomes include the time spent with glucose levels above and below target and other CGM metrics. Safety assessments include the frequency and severity of hypoglycaemic episodes and diabetic ketoacidosis (DKA). In the extension phase, participants have follow-up contacts every 3 months, with the primary endpoint measured over 18 months from the end of the primary phase and compared to sensor augmented pump therapy during that phase. Secondary outcomes, safety, and utility will be assessed similarly.

DETAILED DESCRIPTION:
Purpose of clinical trial:

To determine whether 24/7 automated hybrid closed loop will improve glucose control as measured by time within the target range compared with sensor augmented pump therapy in very young children with T1D.

Study objectives:

The study objective is to evaluate the safety, efficacy and utility of automated hybrid closed loop glucose control in very young children with type 1 diabetes.

1. EFFICACY: The objective is to assess the ability of a hybrid closed loop system to maintain CGM glucose levels within the target range of 3.9 to 10 mmol/l (70 to 180 mg/dl) in comparison with sensor augmented pump therapy in very young children with type 1 diabetes.
2. SAFETY: The objective is to evaluate the safety of closed loop glucose control compared with sensor augmented pump therapy in terms of episodes and severity of hypoglycaemia, frequency of diabetic ketoacidosis (DKA) and nature and severity of other adverse events.
3. UTILITY: The objective is to determine the acceptability and duration of use of the closed loop system in this population.
4. HUMAN FACTORS: The objective is to assess emotional and behavioural characteristics of participants and parents/guardians and their response to the closed loop system and clinical trial using validated surveys and semi-structured qualitative interviews.
5. HEALTH ECONOMICS: The objective is to perform a cost utility analysis to inform reimbursement decision-making.

Participating clinical centres:

1. Addenbrooke's Hospital, Cambridge University Hospital NHS Foundation Trust, Cambridge, UK
2. Leeds Teaching Hospitals NHS Trust, Leeds, UK
3. DECCP, Centre Hospitalier de Luxembourg, Grand Duché de Luxembourg
4. University of Leipzig, Leipzig, Germany
5. Medical University of Graz, Graz, Austria
6. Medical University of Innsbruck, Innsbruck, Austria
7. Medical University of Vienna, Vienna, Austria

Sample Size:

72 participants randomised (8-12 participants per centre). At the primary phase final visit, participants (UK sites only) on sensor-augmented pump therapy as their standard clinical care will be invited to participate in an extension phase of closed loop therapy for a further 18 months.

Maximum duration of study for a subject: 11 months (primary phase). 29 months for participants (UK sites only) opting to participate in 18-month extension phase.

Recruitment:

The subjects will be recruited through paediatric diabetes outpatient clinics at participating clinical centres (see above). Enrolment will target up to 80 (aiming for 8-12 participants per centre) to allow for dropouts during run-in.

Participants (UK sites only) completing the primary phase, who are on sensor-augmented pump therapy as their standard clinical care, will be invited to participate in the extension phase.

Consent:

Written informed consent will be obtained from all parents/guardians and written assent from older children before any study related activities.

Additional written consent will be obtained for the extension phase from all parents/guardians.

Baseline Assessment:

Eligible subjects will undergo a baseline assessment including a blood sample for the measurement of HbA1c. Questionnaires will be completed by parents/guardians.

Pre-Study Training and Run-in:

Training sessions on the use of the study CGM and insulin pump will be provided by the research team. During a 2-4 week run-in period, subjects will use study CGM and insulin pump. For compliance and to assess the ability of the subject to use the study devices safely, at least 8 days of CGM data need to be recorded and safe use of study insulin pump demonstrated during the last 14 days of run-in period. The CGM data will also be used to assess baseline glucose control and may be used for treatment optimization as necessary.

Competency Assessment:

Competency on the use of study insulin pump and study CGM will be evaluated using a competency assessment tool developed by the research team. Training may be repeated if required.

Randomisation:

Eligible subjects will be randomised using randomisation software to the initial use of automated hybrid closed loop glucose system or to sensor augmented pump therapy for 16 weeks with a 1 to 4 week washout period before crossing over to the other study arm.

Automated day and night closed loop insulin delivery (intervention arm)

Participants in the closed loop arm and their caregivers will receive an additional training session covering the use of the closed loop system provided by the research team prior to starting closed loop insulin delivery. During this 1-2 hour session, parents/guardians will operate the system under the supervision of the clinical research team. Competency on the use of closed loop system will be evaluated. Thereafter, subjects and their parents/guardians will use the hybrid closed loop system for 16 weeks at home.

Crossover Assessment:

At the end of the first study arm, a blood sample for the measurement of HbA1c will be taken and weight and height will be measured. Validated surveys evaluating the impact of the devices employed on quality of life, psychosocial function, diabetes management and treatment satisfaction will be completed.

Parents/guardians will be invited to be interviewed to gather feedback on and reactions to their current treatment, the clinical trial, and quality of life changes.

Sensor augmented pump therapy (control arm):

Participants in the sensor augmented pump therapy arm and their caregivers will receive refresher training on key aspects of insulin pump therapy and CGM use.

Subjects and their parents/guardians will continue using sensor augmented pump therapy for 16 weeks at home.

Study contacts:

Participants will be contacted 24h after starting each study arm to ensure there are no concerns regarding the study devices. In between study visits, participants will be contacted by the study team (email/phone) once monthly and 3-monthly in the extension phase, in order to record any adverse events, device deficiencies, and changes in insulin settings, other medical conditions and/or medication.

In case of any problems related to the technical device or diabetes management such as hypo- or hyperglycaemia, subjects will be able to contact a 24-hour telephone helpline to the local research team at any time. The local research team will have access to central 24 hour advice on technical issues.

End of study assessments (primary phase):

A blood sample will be taken for measurement of HbA1c at the end of the study. Height and weight will be recorded. Study devices will be downloaded and returned. Participants will resume usual care using their pre-study insulin pump. Validated surveys evaluating the impact of the devices employed on quality of life, psychosocial function and diabetes management and treatment satisfaction will be completed.

Parents/guardians will be invited to participate in a sleep sub-study prior to the final visit (UK & Luxembourg only).

Parents/guardians will be invited to be interviewed to gather feedback on and reactions to their current treatment, the clinical trial, and quality of life changes.

Extension Phase (UK sites only):

Follow up contacts will be conducted 3-monthly, in line with routine clinic visits, including recording of adverse events, medical history, insulin requirements and HbA1c.

After 18 months from the end of the primary phase, parents/guardians will complete validated questionnaires evaluating the impact of the technology on quality of life, diabetes management, sleep quality and fear of hypoglycaemia. Height and weight will be measured. A blood sample will be taken for measurement of HbA1c at the end of the extension phase

Procedures for safety monitoring during trial:

Standard operating procedures for monitoring and reporting of all adverse events will be in place, including serious adverse events (SAE), serious adverse device effects (SADE) and specific adverse events (AE) such as severe hypoglycaemia.

A data safety and monitoring board (DSMB) will be informed of all serious adverse events and any unanticipated serious adverse device effects that occur during the study and will review compiled adverse event data at periodic intervals.

Criteria for withdrawal of subjects on safety grounds:

A subject/guardian may terminate participation in the study at any time without necessarily giving a reason and without any personal disadvantage. An investigator can stop the participation of a subject after consideration of the benefit/risk ratio. Possible reasons are:

* Serious adverse events
* Non-compliance
* Serious protocol violation
* Decision by the investigator, or the sponsor, that termination is in the subject's best medical interest
* Allergic reaction to insulin

ELIGIBILITY:
Inclusion Criteria:

1. Age between 1 and 7 years (inclusive) (Luxembourg and Austria)
2. Age between 2 and 7 years (inclusive) (Germany and UK)
3. Type 1 diabetes as defined by WHO for at least 6 months [WHO definition: 'The aetiological type named type 1 encompasses the majority of cases which are primarily due to beta-cell destruction, and are prone to ketoacidosis. Type 1 includes those cases attributable to an autoimmune process, as well as those with beta-cell destruction for which neither an aetiology nor a pathogenesis is known (idiopathic). It does not include those forms of beta-cell destruction or failure to which specific causes can be assigned (e.g. cystic fibrosis, mitochondrial defects, etc.).']
4. Insulin pump user (with or without continuous glucose monitoring or flash glucose monitoring system) for at least 3 months, with subject/carer good knowledge of insulin self-adjustment as judged by the investigator
5. On sensor-augmented pump as standard clinical care (extension phase only)
6. Treated with rapid or ultra-rapid acting insulin analogue
7. Subject/carer is willing to perform regular finger-prick blood glucose monitoring, with at least 2 blood glucose measurements taken every day
8. Screening HbA1c ≤ 11% (97mmol/mol) on analysis from local laboratory
9. Willing to wear glucose sensor
10. Willing to wear closed loop system 24/7 during intervention arm
11. The subject/carer is willing to follow study specific instructions
12. The subject/carer is willing to upload pump and CGM data at regular intervals

Exclusion Criteria:

1. Physical or psychological disease likely to interfere with the normal conduct of the study and interpretation of the study results as judged by the investigator
2. Untreated coeliac disease or thyroid disease based on local investigations prior to study enrolment
3. Current treatment with drugs known to interfere with glucose metabolism, e.g. systemic corticosteroids
4. Use of closed loop insulin delivery within the past 2 months
5. Known or suspected allergy to insulin
6. Carer's lack of reliable telephone facility for contact
7. Subject/carer's severe visual impairment
8. Subject/carer's severe hearing impairment
9. Medically documented allergy towards the adhesive (glue) of plasters or subject is unable to tolerate tape adhesive in the area of sensor placement
10. Serious skin diseases (e.g. psoriasis vulgaris, bacterial skin diseases) located in parts of the body which could potentially be used for localisation of the glucose sensor)
11. Sickle cell disease, haemoglobinopathy; or has received red blood cell transfusion or erythropoietin within 3 months prior to time of screening
12. Plan to receive red blood cell transfusion or erythropoietin over the course of study participation
13. Subject/carer not proficient in English (UK, Germany, Austria, Luxembourg) or German (Germany, Austria, Luxembourg) or French (Luxembourg)

    Additional exclusion criteria - Germany only
14. Known microvascular diabetes complications (retinopathy, renal disease, neuropathy)
15. Eating disorders
16. Psychiatric diseases of the parents that would possibly interfere with the ability to comply to study procedures
17. Major needle phobia that would complicate to wear pump catheter and sensor
18. Congenital malformations that would interfere with diabetes treatment (e.g. congenital heart malformations, lung diseases, renal malformations)
19. Growth hormone deficiency
20. Combined Hypopituitarism
21. Down Syndrome (high risk for comorbidity with coeliac disease, autoimmune thyroiditis)
22. Cancer under treatment
23. Current participation in other interventional clinical trials

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2022-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roman Hovorka, Study Director — Wellcome Trust-MRC Institute of Metabolic Science University of Cambridge
Locations (8):
- Austria (3):
  - Medical University of Graz Department of Pediatrics and Adolescent Medicine, Graz
  - Medical University of Innsbruck Department of Pediatrics I, Innsbruck
  - Medical University of Vienna Department of Pediatrics, Vienna
- University of Leipzig Division for Paediatric Diabetology, Leipzig, Germany
- Clinique Pédiatrique de Luxembourg Centre Hospitalier de Luxembourg, Luxembourg, Luxembourg
- United Kingdom (3):
  - University Department of Paediatrics, Cambridge, Cambridgeshire
  - Wellcome Trust-MRC Institute of Metabolic Science University of Cambridge, Cambridge, Cambridgeshire
  - St James's University Hospital, Leeds

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, statistical analysis plan and fully anonymised individual participant data that underlie the results reported in the manuscript will be available 6 months following publication and ending 36 months following manuscript publication to investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose, to achieve aims in the approved proposal. Proposals should be directed to rh347@cam.ac.uk and may be submitted up to 36 months following article publication. To gain access, data requestors will need to sign a data access agreement.
  Fully anonymised data may be shared with third parties (EU or non-EU based) for the purposes of advancing management and treatment of diabetes.
Supporting Information: Study Protocol, SAP
Time Frame: Study protocol, statistical analysis plan and fully anonymised individual participant data that underlie the results reported in the manuscript will be available 6 months following publication and ending 36 months following manuscript publication to investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose, to achieve aims in the approved proposal. Proposals should be directed to rh347@cam.ac.uk and may be submitted up to 36 months following article publication.
Access Criteria: Study protocol, statistical analysis plan and fully anonymised individual participant data that underlie the results reported in the manuscript will be available 6 months following publication and ending 36 months following manuscript publication to investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose, to achieve aims in the approved proposal. Proposals should be directed to rh347@cam.ac.uk and may be submitted up to 36 months following article publication.

REFERENCES:
- [Background] Elleri D, Allen JM, Tauschmann M, El-Khairi R, Benitez-Aguirre P, Acerini CL, Dunger DB, Hovorka R. Feasibility of overnight closed-loop therapy in young children with type 1 diabetes aged 3-6 years: comparison between diluted and standard insulin strength. BMJ Open Diabetes Res Care. 2014 Dec 11;2(1):e000040. doi: 10.1136/bmjdrc-2014-000040. eCollection 2014. PMID 25512874
- [Background] Thabit H, Tauschmann M, Allen JM, Leelarathna L, Hartnell S, Wilinska ME, Acerini CL, Dellweg S, Benesch C, Heinemann L, Mader JK, Holzer M, Kojzar H, Exall J, Yong J, Pichierri J, Barnard KD, Kollman C, Cheng P, Hindmarsh PC, Campbell FM, Arnolds S, Pieber TR, Evans ML, Dunger DB, Hovorka R. Home Use of an Artificial Beta Cell in Type 1 Diabetes. N Engl J Med. 2015 Nov 26;373(22):2129-2140. doi: 10.1056/NEJMoa1509351. Epub 2015 Sep 17. PMID 26379095
- [Background] Tauschmann M, Allen JM, Wilinska ME, Thabit H, Stewart Z, Cheng P, Kollman C, Acerini CL, Dunger DB, Hovorka R. Day-and-Night Hybrid Closed-Loop Insulin Delivery in Adolescents With Type 1 Diabetes: A Free-Living, Randomized Clinical Trial. Diabetes Care. 2016 Jul;39(7):1168-74. doi: 10.2337/dc15-2078. Epub 2016 Jan 6. PMID 26740634
- [Background] Tauschmann M, Allen JM, Wilinska ME, Thabit H, Acerini CL, Dunger DB, Hovorka R. Home Use of Day-and-Night Hybrid Closed-Loop Insulin Delivery in Suboptimally Controlled Adolescents With Type 1 Diabetes: A 3-Week, Free-Living, Randomized Crossover Trial. Diabetes Care. 2016 Nov;39(11):2019-2025. doi: 10.2337/dc16-1094. Epub 2016 Sep 9. PMID 27612500
- [Derived] Ware J, Allen JM, Boughton CK, Wilinska ME, Hartnell S, Thankamony A, de Beaufort C, Schierloh U, Frohlich-Reiterer E, Mader JK, Kapellen TM, Rami-Merhar B, Tauschmann M, Nagl K, Hofer SE, Campbell FM, Yong J, Hood KK, Lawton J, Roze S, Sibayan J, Bocchino LE, Kollman C, Hovorka R; KidsAP Consortium. Randomized Trial of Closed-Loop Control in Very Young Children with Type 1 Diabetes. N Engl J Med. 2022 Jan 20;386(3):209-219. doi: 10.1056/NEJMoa2111673. PMID 35045227
- [Derived] Fuchs J, Allen JM, Boughton CK, Wilinska ME, Thankamony A, de Beaufort C, Campbell F, Yong J, Froehlich-Reiterer E, Mader JK, Hofer SE, Kapellen TM, Rami-Merhar B, Tauschmann M, Hood K, Kimbell B, Lawton J, Roze S, Sibayan J, Cohen N, Hovorka R; KidsAP Consortium. Assessing the efficacy, safety and utility of closed-loop insulin delivery compared with sensor-augmented pump therapy in very young children with type 1 diabetes (KidsAP02 study): an open-label, multicentre, multinational, randomised cross-over study protocol. BMJ Open. 2021 Feb 12;11(2):e042790. doi: 10.1136/bmjopen-2020-042790. PMID 33579766

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 81 participants were enrolled between 17 May 201 9 and 16 June 2020 at 7 paediatric diabetes centres in the UK, Luxembourg, Austria and Germany.
Pre-assignment Details: 74 out of 81 enrolled participants were randomised. Of those not randomised two were withdrawn by the site due to safety concerns and five chose not to continue with the study.
Groups:
- Closed-loop Insulin Delivery (Intervention), Then Sensor-augmented Pump Therapy (Control): Unsupervised home use of day and night automated hybrid closed loop insulin delivery system for 16 weeks.
  Intervention: Device: CamAPS FX
  CamAPS FX: CamAPS FX closed loop system comprises:
  * Dana insulin pump (Diabecare, Sooil, Seoul, South Korea)
  * Dexcom G6 real-time CGM sensor (Dexcom, Northridge, CA, USA)
  * An Android smartphone hosting CamAPS FX app with the Cambridge model predictive control algorithm and communicating wirelessly with the insulin pump and glucose sensor
  * Cloud upload system to monitor CGM/insulin data
  After a washout period of 1-4 weeks, use of sensor-augmented pump therapy for 16 weeks.
  Sensor augmented therapy: Study insulin pump and study CGM.
- Sensor Augmented Pump Therapy (Control), Then Closed-loop Insulin Delivery (Intervention): Sensor augmented pump therapy for 16 weeks.
  Sensor augmented therapy: Study insulin pump and study CGM.
  After a washout period of 1-4 weeks, unsupervised home use of day and night automated hybrid closed loop insulin delivery system for 16 weeks.
  Intervention: Device: CamAPS FX
  CamAPS FX: CamAPS FX closed loop system comprises:
  * Dana insulin pump (Diabecare, Sooil, Seoul, South Korea)
  * Dexcom G6 real-time CGM sensor (Dexcom, Northridge, CA, USA)
  * An Android smartphone hosting CamAPS FX app with the Cambridge model predictive control algorithm and communicating wirelessly with the insulin pump and glucose sensor
  * Cloud upload system to monitor CGM/insulin data
Period: Period 1
Arm/Group | Closed-loop Insulin Delivery (Intervention), Then Sensor-augmented Pump Therapy (Control) | Sensor Augmented Pump Therapy (Control), Then Closed-loop Insulin Delivery (Intervention)
Started | 39 | 35
Completed | 39 | 34
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Washout
Arm/Group | Closed-loop Insulin Delivery (Intervention), Then Sensor-augmented Pump Therapy (Control) | Sensor Augmented Pump Therapy (Control), Then Closed-loop Insulin Delivery (Intervention)
Started | 39 | 34
Completed | 39 | 34
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Closed-loop Insulin Delivery (Intervention), Then Sensor-augmented Pump Therapy (Control) | Sensor Augmented Pump Therapy (Control), Then Closed-loop Insulin Delivery (Intervention)
Started | 39 | 34
Completed | 39 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Closed-loop Insulin Delivery First, Then Sensor-augmented Pump Therapy: Unsupervised home use of day and night automated hybrid closed loop insulin delivery system for 16 weeks.
  Intervention: Device: CamAPS FX
  CamAPS FX: CamAPS FX closed loop system comprises:
  * Dana insulin pump (Diabecare, Sooil, Seoul, South Korea)
  * Dexcom G6 real-time CGM sensor (Dexcom, Northridge, CA, USA)
  * An Android smartphone hosting CamAPS FX app with the Cambridge model predictive control algorithm and communicating wirelessly with the insulin pump and glucose sensor
  * Cloud upload system to monitor CGM/insulin data
  Following a 1-4 week washout period, use of sensor-augmented pump therapy for 16 weeks.
  Sensor augmented therapy: Study insulin pump and study CGM.
- Sensor Augmented Pump Therapy First, Then Closed-loop Insulin Delivery: Sensor augmented pump therapy for 16 weeks.
  Sensor augmented therapy: Study insulin pump and study CGM.
  Following a 1-4 week washout period, unsupervised home use of day and night automated hybrid closed loop insulin delivery system for 16 weeks.
  Intervention: Device: CamAPS FX
  CamAPS FX: CamAPS FX closed loop system comprises:
  * Dana insulin pump (Diabecare, Sooil, Seoul, South Korea)
  * Dexcom G6 real-time CGM sensor (Dexcom, Northridge, CA, USA)
  * An Android smartphone hosting CamAPS FX app with the Cambridge model predictive control algorithm and communicating wirelessly with the insulin pump and glucose sensor
  * Cloud upload system to monitor CGM/insulin data
- Total: Total of all reporting groups
Arm/Group | Closed-loop Insulin Delivery First, Then Sensor-augmented Pump Therapy | Sensor Augmented Pump Therapy First, Then Closed-loop Insulin Delivery | Total
Number analyzed (Participants) | 39 | 35 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.6 (1.4) | 5.6 (1.7) | 5.6 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 10 | 31
  Male | 18 | 25 | 43
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 34 | 32 | 66
  Black | 2 | 0 | 2
  Asian | 1 | 1 | 2
  Multiple | 2 | 2 | 4
Duration of diabetes [Mean (Standard Deviation); unit: years] | 2.5 (1.7) | 2.7 (1.9) | 2.6 (1.8)
Continuous Glucose Monitor Use [Count of Participants; unit: Participants]
  Current | 35 | 32 | 67
  In past but not current | 0 | 1 | 1
  Never | 4 | 2 | 6
BMI percentile (age- and sex-adjusted) [Mean (Standard Deviation); unit: percentile] | 67.3 (23.2) | 71.1 (24.6) | 69.1 (23.8)
HbA1c at screening [Mean (Standard Deviation); unit: % of glucose linked to haemoglobin] | 7.3 (0.7) | 7.4 (0.6) | 7.3 (0.7)
HbA1c [Mean (Standard Deviation); unit: mmol/mol] | 56.3 (7.4) | 57 (7.1) | 56.6 (7.2)
Percent of time in glucose range of 70-180 mg/dl [Mean (Standard Deviation); unit: %] | 61.5 (9.5) | 60.8 (10.9) | 61.2 (10.1)
Continuous glucose monitoring metrics at baseline [Median (Inter-Quartile Range); unit: percentage of time]
  Median percent of time with sensor glucose >180mg/dL (%) | 32.2 [24.0 to 42.7] | 36.7 [21.6 to 41.8] | 34.4 [24.0 to 42.2]
  Median percent of time with sensor glucose >300mg/dL (%) | 3.4 [2.0 to 7.9] | 3.8 [1.2 to 8.5] | 3.7 [1.8 to 7.9]
  Median percent of time with sensor glucose <70mg/dL (%) | 4.5 [2.4 to 6.7] | 3.9 [2.0 to 7.4] | 4.4 [2.3 to 7.0]
  Median percent of time with sensor glucose <54mg/dL (%) | 0.8 [0.2 to 1.8] | 0.6 [0.3 to 1.4] | 0.7 [0.3 to 1.6]
Mean sensor glucose [Mean (Standard Deviation); unit: mg/dL] | 162.1 (21.6) | 162.1 (21.6) | 162.1 (21.6)
Standard deviation of glucose [Median (Inter-Quartile Range); unit: mg/dL] | 66.6 [59.4 to 73.9] | 66.6 [55.8 to 77.5] | 66.6 [57.6 to 73.9]
Coefficient of variation of glucose [Median (Inter-Quartile Range); unit: %] | 42.4 [36.9 to 45.0] | 41.1 [36.6 to 43.9] | 41.6 [36.6 to 43.9]
Median total daily insulin (U/kg/day) [Median (Inter-Quartile Range); unit: Units/kg/day] | 0.76 [0.67 to 0.83] | 0.77 [0.69 to 0.86] | 0.76 [0.67 to 0.85]

OUTCOME MEASURES:

1. Primary Outcome: Time in Target (3.9 to 10.0 mmol/l) (70 to 180 mg/dl)
Description: Between group difference in time spent with sensor glucose levels between 3.9 to 10.0 mmol/l (70 to 180 mg/dl) during the 4 months intervention period.
Time Frame: 16-week home stay
Measure: Mean (Standard Deviation); unit: Percent of time spent in target range
Groups:
- Closed-loop Period: Unsupervised home use of day and night automated hybrid closed loop insulin delivery system over 16 weeks.
  Intervention: Device: CamAPS FX
  CamAPS FX: CamAPS FX closed loop system comprises:
  * Dana insulin pump (Diabecare, Sooil, Seoul, South Korea)
  * Dexcom G6 real-time CGM sensor (Dexcom, Northridge, CA, USA)
  * An Android smartphone hosting CamAPS FX app with the Cambridge model predictive control algorithm and communicating wirelessly with the insulin pump and glucose sensor
  * Cloud upload system to monitor CGM/insulin data
- Sensor-augmented Pump Period: Sensor augmented pump therapy over 16 weeks.
  Sensor augmented therapy: Study insulin pump and study CGM.
Arm/Group | Closed-loop Period | Sensor-augmented Pump Period
Number analyzed (Participants) | 73 | 74
Percent of time spent in target range | 71.6 (5.9) | 62.9 (9.0)
Statistical Analysis 1: Comparison: Closed-loop Period vs Sensor-augmented Pump Period; Test type: Superiority; p < 0.001, Regression, Linear; Mean Difference (Final Values) = 8.7, 95% CI 2-sided [7.4 to 9.9] — The mean adjusted differences are based on a linear mixed model with adjustment for repeated participant measures, with period as a fixed effect and trial site as a random effect; the model also accounted for the baseline values

2. Secondary Outcome: Key Endpoint: Time Spent Above Target Glucose (10.0 mmol/l) (180 mg/dl)
Description: Percentage of time spent with sensor glucose readings above target glucose (10.0mmol/l) (180mg/dl)
Time Frame: 16-week home stay
Measure: Median (Inter-Quartile Range); unit: Percent of time spent
Arm/Group | Closed-loop Period | Sensor-augmented Pump Period
Number analyzed (Participants) | 73 | 74
Percent of time spent | 22.9 [19.3 to 27.3] | 31.7 [23.4 to 40.1]
Statistical Analysis 1: Comparison: Closed-loop Period vs Sensor-augmented Pump Period; Test type: Superiority; p < 0.001, Regression, Linear — The primary and key secondary end points were tested in hierarchy (Time in range, time >180mg/dL, HbA1c, mean glucose, time <70mg/dL) to control the type 1 error with the use of the fixed-sequence method; Mean Difference (Final Values) = -8.5, 95% CI 2-sided [-9.9 to -7.1] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Key Endpoint: HbA1c
Description: HbA1c is measured in % as per NGSP
Time Frame: 16-week home stay
Measure: Mean (Standard Deviation); unit: % of glucose linked to haemoglobin molec
Arm/Group | Closed-loop Period | Sensor-augmented Pump Period
Number analyzed (Participants) | 73 | 74
% of glucose linked to haemoglobin molec | 6.6 (0.6) | 7.0 (0.7)
Statistical Analysis 1: Comparison: Closed-loop Period vs Sensor-augmented Pump Period; Test type: Superiority; p < 0.001, Regression, Linear — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.5 to -0.3] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Key Endpoint: HbA1c
Description: HbA1c, measured using standardized, validated assays, serves as an indicator of long-term glycemic control, reflecting the average blood glucose levels over approximately 3 months.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | Closed-loop Period | Sensor-augmented Pump Period
Number analyzed (Participants) | 73 | 74
mmol/mol | 49.0 (5.9) | 52.8 (7.2)
Statistical Analysis 1: Comparison: Closed-loop Period vs Sensor-augmented Pump Period; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -3.9, 95% CI 2-sided [-4.9 to -2.9]

5. Secondary Outcome: Key Endpoint: Mean Sensor Glucose
Description: Mean sensor glucose is calculated from CGM readings over the study period to reflect overall glycemic control.
Time Frame: 16-week home stay
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Closed-loop Period | Sensor-augmented Pump Period
Number analyzed (Participants) | 73 | 74
mg/dL | 145.8 (11.8) | 158.1 (18.5)
Statistical Analysis 1: Comparison: Closed-loop Period vs Sensor-augmented Pump Period; Test type: Superiority; p < 0.001, Regression, Linear — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -12.3, 95% CI 2-sided [-14.8 to -9.8] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Key Endpoint: Time Spent Below Target Glucose (3.9 mmol/l) (70 mg/dl)
Description: Percentage of time spent with sensor glucose readings below target glucose (3.9mmol/l)(70mg/dl)
Time Frame: 16-week home stay
Measure: Median (Inter-Quartile Range); unit: Percent of time spent
Arm/Group | Closed-loop Period | Sensor-augmented Pump Period
Number analyzed (Participants) | 73 | 74
Percent of time spent | 4.9 [3.3 to 6.7] | 4.5 [2.9 to 7.3]
Statistical Analysis 1: Comparison: Closed-loop Period vs Sensor-augmented Pump Period; Test type: Superiority; p = 0.74, Regression, Linear — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.4 to 0.5]

7. Secondary Outcome: Standard Deviation
Description: Standard deviation of sensor glucose levels
Time Frame: 16-week home stay
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Closed-loop Period | Sensor-augmented Pump Period
Number analyzed (Participants) | 73 | 74
mg/dL | 58.6 [53.7 to 64.4] | 64.2 [58.1 to 71.9]
Statistical Analysis 1: Comparison: Closed-loop Period vs Sensor-augmented Pump Period; Test type: Superiority — The mean adjusted differences are based on a linear mixed model with adjustment for repeated participant measures, with period as a fixed effect and trial site as a random effect; the model also accounted for the baseline values; Mean Difference (Final Values) = -6.2, 95% CI 2-sided [-7.6 to -4.8] — Confidence intervals for the secondary end points were adjusted for multiple comparisons with the use of the Benjamini-Hochberg procedure to control the false discovery rate

8. Secondary Outcome: Coefficient of Variation (Percentage) of Glucose Levels
Description: Coefficient of variation (percentage) of sensor glucose levels
Time Frame: 16-week home stay
Measure: Median (Inter-Quartile Range); unit: Percent
Arm/Group | Closed-loop Period | Sensor-augmented Pump Period
Number analyzed (Participants) | 73 | 74
Percent | 41 [39 to 43] | 41 [38 to 44]
Statistical Analysis 1: Comparison: Closed-loop Period vs Sensor-augmented Pump Period; Test type: Superiority — The mean adjusted differences are based on a linear mixed model with adjustment for repeated participant measures, with period as a fixed effect and trial site as a random effect; the model also accounted for the baseline values. Differences in percents are shown in percentage points; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-1.5 to 0.05] — [estimate comment as in outcome 7, analysis 1]

9. Secondary Outcome: Time With Glucose Levels <3.0 mmol/l (54 mg/dl)
Description: Percentage of time spent with glucose levels < 3.0mmol/l (54 mg/dl)
Time Frame: 16-week home stay
Measure: Median (Inter-Quartile Range); unit: Percent of time spent
Arm/Group | Closed-loop Period | Sensor-augmented Pump Period
Number analyzed (Participants) | 73 | 74
Percent of time spent | 1.0 [0.6 to 1.4] | 0.9 [0.4 to 1.6]
Statistical Analysis 1: Comparison: Closed-loop Period vs Sensor-augmented Pump Period; Test type: Superiority; The mean adjusted differences are based on a linear mixed model with adjustment for repeated participant measures, with period as a fixed effect and trial site as a random effect; the model also accounted for the baseline values; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.1 to 0.1] — [estimate comment as in outcome 7, analysis 1]

10. Secondary Outcome: Time With Glucose Levels in Significant Hyperglycaemia (Glucose Levels > 16.7 mmol/l) (300 mg/dl)
Description: Percentage of time spent with glucose levels in significant hyperglycaemia (glucose levels > 16.7mmol/l) (300mg/dl)
Time Frame: 16-week home stay
Measure: Median (Inter-Quartile Range); unit: Percent of time spent
Arm/Group | Closed-loop Period | Sensor-augmented Pump Period
Number analyzed (Participants) | 73 | 74
Percent of time spent | 2.0 [1.2 to 3.1] | 3.1 [1.3 to 5.7]
Statistical Analysis 1: Comparison: Closed-loop Period vs Sensor-augmented Pump Period; Test type: Superiority — [test comment as in outcome 7, analysis 1]; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-1.6 to -0.6] — [estimate comment as in outcome 7, analysis 1]

11. Secondary Outcome: AUC of Glucose Below 3.5 mmol/l (63 mg/dl)
Description: Area under the curve of sensor glucose readings below 3.5mmol/l (63mg/dl). Glucose AUC was calculated by trapezoidal approximation of sensor glucose levels.
Time Frame: 16-week home stay
Measure: Median (Inter-Quartile Range); unit: mg*min/dL
Arm/Group | Closed-loop Period | Sensor-augmented Pump Period
Number analyzed (Participants) | 73 | 74
mg*min/dL | 0.1 [0.0 to 0.1] | 0.1 [0.0 to 0.1]
Statistical Analysis 1: Comparison: Closed-loop Period vs Sensor-augmented Pump Period; Test type: Non-Inferiority — [test comment as in outcome 7, analysis 1]; Mean Difference (Final Values) = 0.002, 95% CI 2-sided [-0.006 to 0.009] — [estimate comment as in outcome 7, analysis 1]

12. Secondary Outcome: BMI SDS
Description: BMI Standard Deviation Score
Time Frame: 16-week home stay
Measure: Mean (Standard Deviation); unit: Percentile
Arm/Group | Closed-loop Period | Sensor-augmented Pump Period
Number analyzed (Participants) | 65 | 68
Percentile | 71 (23) | 70 (26)
Statistical Analysis 1: Comparison: Closed-loop Period vs Sensor-augmented Pump Period; Test type: Superiority; p = 0.75, Regression, Linear; Based on a longitudinal model adjusting for baseline value and period as fixed effects. The model accounts for correlated data from the same subject; Mean Difference (Final Values) = 0.004, 95% CI 2-sided [-0.02 to 0.03]

13. Secondary Outcome: Total, Basal, and Bolus Insulin Dose
Description: Median daily total, basal and bolus insulin use
Time Frame: 16-week home stay
Measure: Median (Inter-Quartile Range); unit: Units/day
Arm/Group | Closed-loop Period | Sensor-augmented Pump Period
Number analyzed (Participants) | 73 | 74
Units/day
  Total daily insulin use | 16.9 [13.2 to 21.5] | 17.6 [13.6 to 20.3]
  Total daily basal insulin use | 8.0 [5.8 to 10.9] | 5.7 [4.0 to 6.9]
  Total daily bolus insulin use | 8.6 [6.9 to 10.6] | 11.0 [9.1 to 13.5]
Statistical Analysis 1: Comparison: Closed-loop Period vs Sensor-augmented Pump Period; Test type: Superiority — [test comment as in outcome 7, analysis 1]; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-0.1 to 0.8] — (For total daily insulin use) Confidence intervals for the secondary end points were adjusted for multiple comparisons with the use of the Benjamini-Hochberg procedure to control the false discovery rate

14. Secondary Outcome: Number of Episodes of Severe Hypoglycaemia
Description: This outcome measure records the total number of severe hypoglycaemic episodes-defined as events requiring external assistance-experienced during the study period. Episodes are captured through patient records and clinical confirmation.
Time Frame: 16-week home stay
Measure: Number; unit: number of events
Arm/Group | Closed-loop Period | Sensor-augmented Pump Period
Number analyzed (Participants) | 73 | 74
number of events | 1 | 0

15. Secondary Outcome: Number of Subjects Experiencing Severe Hypoglycaemia
Description: Count of subjects with at least one severe hypoglycaemic event during the study. Severe events are defined as episodes requiring external assistance.
Time Frame: 16-week home stay
Measure: Count of Participants; unit: Participants
Arm/Group | Closed-loop Period | Sensor-augmented Pump Period
Number analyzed (Participants) | 73 | 74
Participants | 1 | 0

16. Secondary Outcome: Frequency of Diabetic Ketoacidosis
Description: The incidence of diabetic ketoacidosis (DKA) episodes will be recorded as the number of confirmed events during the study
Time Frame: 16-week home stay
Measure: Count of Participants; unit: Participants
Arm/Group | Closed-loop Period | Sensor-augmented Pump Period
Number analyzed (Participants) | 73 | 74
Participants | 0 | 0

17. Secondary Outcome: Frequency and Nature of Other Adverse Events
Description: The frequency and nature of other adverse events will be recorded throughout the study. All events not directly linked to the intervention will be documented, detailing their onset, duration, severity, and potential relation to the treatment.
Time Frame: 16-week home stay
Measure: Count of Participants; unit: Participants
Arm/Group | Closed-loop Period | Sensor-augmented Pump Period
Number analyzed (Participants) | 73 | 74
Participants
  Number of participants with no adverse events | 53 | 56
  Number of participants with one adverse event | 15 | 12
  Number of participants with two or more adverse events | 5 | 6

18. Secondary Outcome: Percentage of Time of CGM Availability
Description: This outcome assesses the percentage of time the continuous glucose monitoring (CGM) system is active and delivering valid data.
Time Frame: 16-week home stay
Measure: Median (Inter-Quartile Range); unit: Time using CGM (%)
Arm/Group | Closed-loop Period | Sensor-augmented Pump Period
Number analyzed (Participants) | 73 | 74
Time using CGM (%) | 99 [99 to 100] | 99 [99 to 100]

19. Secondary Outcome: Percentage of Time of Closed-loop Operation
Description: This outcome measure determines the percentage of the total study period during which the closed-loop insulin delivery system operates as intended.
Time Frame: 16-week home stay
Measure: Median (Inter-Quartile Range); unit: Time using closed-loop (%)
Arm/Group | Closed-loop Period
Number analyzed (Participants) | 73
Time using closed-loop (%) | 95 [92 to 97]

20. Secondary Outcome: Frequency and Nature of Other Serious Adverse Events
Description: Frequency and nature of other serious adverse events will be documented, including type, severity, and potential treatment association.
Time Frame: 16-week home stay
Measure: Count of Participants; unit: Participants
Arm/Group | Closed-loop Period | Sensor-augmented Pump Period
Number analyzed (Participants) | 73 | 74
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Over both 16-week study periods (total 32 weeks).
Description: Severe hypoglycaemia was defined as per ISPAD guidance: If the event requires assistance of another person due to altered consciousness to actively administer carbohydrate, glucagon, or other resuscitative actions. This means that the subject is impaired cognitively to the point that he/she is unable to treat him- or herself, is unable to verbalize his or her needs, is incoherent, disoriented, and/or combative, or experiences seizure or coma.
Arm/Group | Closed-loop Period | Sensor-augmented Pump Period
All-Cause Mortality (participants affected / at risk) | 0/73 | 0/74
Serious Adverse Events (participants affected / at risk) | 1/73 | 1/74
Other Adverse Events (participants affected / at risk) | 20/73 | 18/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Closed-loop Period (N=73) | Sensor-augmented Pump Period (N=74)
Severe hypoglycaemia event (Endocrine disorders) | 1 (1) | 0 (0) — The parents had set the nocturnal personal glucose target to 80 mg/dL. Before the severe hypoglycemia event, an audio alarm was issued overnight every 5 minutes for 3 hours. Alarms were acknowledged by the parents, but no hypo treatment was given.
Other serious adverse event. (Gastrointestinal disorders) | 0 (0) | 1 (1) — Hospital admission for gastroenteritis
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Closed-loop Period (N=73) | Sensor-augmented Pump Period (N=74)
Hyperglycaemia (Endocrine disorders) | 2 (2) | 6 (10)
Infection (Cold, UTI, D&V, fever) (Infections and infestations) | 16 (24) | 11 (16)
Head injury (Nervous system disorders) | 0 (0) | 1 (1)
Diabetes related (Product Issues) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-05): https://cdn.clinicaltrials.gov/large-docs/27/NCT03784027/Prot_SAP_000.pdf